CLINICAL TRIAL: NCT03995381
Title: Using Decision Aids to Reducing Decision Conflict in Angiography Patients for Choosing Hemostasis: A Randomized Controlled Trial
Brief Title: Using Decision Aids to Reducing Decision Conflict in Angiography Patients for Choosing Hemostasis
Acronym: N201902036
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201902036
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-06

CONDITIONS: Haemostatic Adverse Reaction
Keywords: Haemostasis
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAs group (Experimental): Shared decision making using decision aids
  Interventions: Other: Decision aids
- Control group (No Intervention): Standard oral explanation guided with booklets

INTERVENTIONS:
Other: Decision aids — Shared decision making with decision aids
  Arms: DAs group

SUMMARY:
Vascular closure device, hemostatic bandage and manual compression can achieve hemostasis after angiographic examination. These three methods of hemostasis changed the rate of hemostasis, early ambulation, hematoma , hemostasis failure rate, and expense. Therefore, shared decision making (SDM) is necessary to aid patients to choose hemostasis.The investigators have developed a decision aids (DA) and planned a randomized controlled trial (RCT) to evaluate its impact on angiographic patients. The measurements include a battery of interview-based questionnaires and evaluations of decision conflicts. The investigators expect the DAs would benefit the intervention group in the aspects of knowledge, communication and choice conflicts.during and after thier Hemostasis procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who needs an angiographic examination or treatment.
* Patients with angiographic indications
* Patients who were able to give consent and complete the interview

Exclusion Criteria:

* The angiographic procedure uses patients with a catheter size more than 7fr.
* Patients in critical situations requiring urgent treatment
* Patients had cognitive impairment
* Patients were physically unfit to be interviewed
* Patients were non-Mandarin or -Taiwanese

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | 1 hour before Angiography
  Total score of decisional conflict scale

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No